CLINICAL TRIAL: NCT07250607
Title: Extreme Phenotypes to Identify the Patients With Type 2 Diabetes Who Are Susceptible or Resistant to Complications and to Reveal the Mechanisms
Brief Title: Extreme Phenotypes to Identify Susceptibility of Patients Living With Type 2 to Diabetes Related Complications
Acronym: EXTREME-T2D
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Prof., Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: EXTREME-T2D phase 1
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diabete Type 2; Diabetes Complications
Keywords: microvascular complications; macrovascular complications; Type 2 Diabetes Mellitus; Cardiovascular diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subject with Highest susceptibility to complications (HS-DRC): Subjects showing a number of diabetes related complication higher than expected compared with other subject with similar disease duration and glycemic control
- Subject with lowest susceptibility to complications (LS-DRC): Subjects showing a number of diabetes related complication lower than expected compared with other subject with similar disease duration and glycemic control
- Subject with moderate susceptibility to complications (MS-DRC or control gtoup): Subjects showing a number of diabetes related complication that is expected for their disease duration and glycemic control according to the DRC distribution in the general T2D population

SUMMARY:
The goal of this observational study is to learn more about the diverse susceptibility to micro and macrovascular complications in individuals living with Type 2 Diabetes (T2D).

The main questions of the study are:

* Is the chronic exposure to hyperglycemia the only determinant of diverse susceptibility to diabetes related complications (DRC) across the T2D population?
* Is it possible to develop a reliable tool to identify patients at different susceptibility to DRC?
* Is it possible to predict DRC susceptibility through biomarkers in the field of inflammation, hormonal signaling or non-coding circulating nucleotides.

People living with T2D and well screened for complications according to the international recommendations (American Diabetes Association/European Society for the study of Diabetes) will be included in the survey collecting information about chronic exposure to hyperglycemia (diabetes duration + glycemic control) and incidence and severity of each macro and microvascular complication.

Based on the survey result, a clinical score will be proposed to distinguish patient at different susceptibility to complications.

Then, patients with extreme phenotypes of susceptibility (i.e. those with highest susceptibility for their short exposure to hyperglycemia vs those with lowest susceptibility to complication for their long exposure to hyperglycemia) will be recruited to perform a blood drawn and investigate whether preidentified potential biomarkers could describe the diverse susceptibility to DRC by showing a significant gradient between groups.

DETAILED DESCRIPTION:
The incidence of diabetes related complications (DRC) in individuals living with type 2 diabetes (T2D) is known to depend on exposure to disease and risk factor control, but it displays a large interindividual variability. In this observational trial we will explore the feasibility to develop a method to estimate the degree of susceptibility to DRC in any single patient living with T2D, based on a standardized clinical assessment.

The study will consist in a systematic review of the clinical records of patients with T2D, referring 4 different diabetes clinics in Italy and Greece, who undergo a regular follow up and a complete assessment for DRC pertaining to 3 major macrovascular (coronary, cerebrovascular and peripheral) and 3 major microvascular (retina, kidney and peripheral nerves) districts. The diseases will be classified as a overt or subclinical in relation to their clinical significance. The clinical criteria for the classification will be standardized across the centers.

The final population (target= 1000 patients) will be then used to test the ability of a score (DRC score) to categorize each individual in a specific subgroup for DRC burden, that reflects the DRC susceptibility.

The DRC score has been designed by a consensus of expert, and calculated as the sum of each overt (3 points) and subclinical (1 point) micro- and macrovascular complication.

By applying the DRC score to the general T2D population referring to the study centers, we expect to select 120 subject with high susceptibility to complications (HS-DRC) and 120 subject with low susceptibility to complications (LS-DRC). These subject will undergo a blood drawn and full characterization of risk factors to test the ability of these biomarkers in predicting complications occurrence, when compared with a control population of T2D patients with moderate susceptibility to complications.

The potential biomarkers identified after a systematic review of the literature will be:

Environmental and lifestyle modulators: Smoke load; Fluctuations of body mass index (BMI), HbA1C, Blood pressure, lipid profile, kidney function; physical activity; diet quality; sleep quality.

Biological modulators of damage: IGF1, insulin, testosterone, leptin, glucagon; circulating non-coding microRNA related to diabetes complications.

Biological transducers of damage: hsCRP (high sensitivity C reactive proteine), interleukin-6, -1beta and -18, tumor necrosis factor alfa, tumor growth factor beta; carboxyl methyl-lysine, pentosidine; total antioxidant capacity, 3-nitrotyrosines, malondialdehyde.

Will be selected as biomarkers with predictive potential for DRC susceptibility all biomarkers showing a clear and unidirectional gradient between the two extreme phenotypes selected by using the proposed DRC score.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Age 40-80 years old
* Comprehensive screening for DRC within 24 months from the inclusion in the survey.

Exclusion Criteria:

Diagnosis of forms of diabetes other than T2D

* Any chronic inflammatory diseases or active cancer
* Significant liver disfunction (cirrhosis, AST/ALT > 3-fold normality range, total bilirubin > 1,5-fold normal range w/o Gilbert syndrome)
* Any other life expectancy-changing systemic disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Either sex, age between 40 and 80 years old. Diagnosed Type 2 diabetes (proven of exclusion of other forms diabetes if required by the PI) followed up regularly for T2D and with a comprehensive screening for complications including data on coronary, cerevrovascular and peripheral artery disease, and informations about chronic kidney, retinopathy and neuropathy diseases related to diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Diabetes Related Complications. | through study completion, an average of 12 months
  to measure the incidence and intensity of each included micro and macrovascular complication

SECONDARY OUTCOMES:
DRC score | Through study completion, an average of 12 months
  To test the power of the designed score in categorizing patients for the diverse susceptibility to DRC
Biomarkers | through study completion, an average of 12 months
  To select biomarkers for DRC susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, MD, Principal Investigator — University of Pisa
Locations (3):
- Italy (3):
  - Policlinico Consorziale di Bari, Bari, BA
  - Azienda Rilievo Nazionale Alta Specialità (ARNAS) Garibaldi, Catania, CT
  - Azienda Ospedaliero Universitaria Pisana, Pisa, PI

IPD SHARING:
Plan to Share IPD: Undecided